CLINICAL TRIAL: NCT06865703
Title: Efficacy of Different Osteopathic Manipulative Techniques Combined With Diaphragmatic Release in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy of Osteopathic Manipulative Techniques in Patients With Chronic Obstructive Pulmonary Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Shimaa Mokhtar, Physiotherapist, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Osteopathic Techniques in COPD
Record Dates: First submitted 2025-02-24; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Copd
Keywords: diaphragmatic release; rib raising; thoracic lymphatic pump
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: moderate to severe copd
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Other): Combination between rib raising and diaphragmatic release technique
  Interventions: Other: diaphragmatic release technique; Other: rib raising technique in group A
- group B (Other): combination between thoracic lymphatic pump and diaphragmatic release technique
  Interventions: Other: diaphragmatic release technique; Other: THORACIC LYMPHATIC PUMP TECHNIGUE
- group C (control group) (Other): Diaphragmatic release technique (control group)
  Interventions: Other: diaphragmatic release technique

INTERVENTIONS:
Other: diaphragmatic release technique — The participant lay in the supine position and the therapist stood at the participant's head, the therapist passed his hands (the hypothenar and the lateral 3 fingers) under the costal cartilage of the seventh to the tenth ribs bilaterally, with the therapist's forearm aligned up toward the subject's shoulder. Then, the therapist quietly drew the diaphragm in and upward during the inspiratory phase. The therapist then went deeply with both hands toward the inner costal margin during the expiratory phase to resist the rebounding movement of the thoracic cage. The depth of this manual contact was progressively increased in subsequent respiratory cycles. The maneuver was repeated in 4 sets, each of which consisted of 5 deep breaths with 2-min intervals in between if needed
Other: rib raising technique in group A — • The patient is in supine position and therapist hand under the thorax The fingertips take up contact with the angular costae and move it up and in lateral traction and maintained and this will repeated until all ribs on the side are mobilized. This movement will be repeated several times until perceives an improvement in the rib flexibility
  Arms: group A
Other: THORACIC LYMPHATIC PUMP TECHNIGUE — * Patient in the supine position and therapist will stand the participant's head, facing The therapist places the thenar eminence of each hand to the pectoral region and infra clavicular and the other fingers were spread around the thoracic cage and angled toward the body's side to create consistent, compressive force across the thoracic cage The participant was then allowed to breathe in deeply and breath out. The therapist slowly reduced the compressive force and withdrew the participant.
  * During breath out rhythmic oscillatory compression in the posterior and caudal direction was applied to the chest wall.
  * By the end of the expiratory phase, the compressive force was maintained, and ask to take another deep breath. In this way, the participant encountered some resistance equivalent to the chest-wall movement during inspiration. The maneuver was repeated for 5 respiratory cycles, then hands to allow for full inspiration.
  Arms: group B

SUMMARY:
This study will test the efficiency of rib rising technique and thoracic lymphatic pump technique combining with manual diaphragmatic release technique in patients with chronic obstructive pulmonary disease

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a complex and constantly evolving pathology which is characterized by a progressive and constant limitation of the available air volume.

The Global Initiative for Chronic Obstructive Lung Disease (GOLD) identifies COPD as: a common, preventable and treatable disease that is characterized by persistent respiratory symptoms and airflow limitation that is due to airway and/or alveolar abnormalities usually caused by significant exposure to noxious particles or gases.

COPD could become the third leading cause of death for the population by 2030.

Exacerbation 0f COPD leads to hospital admission, high mortality and a decline in the ability to carry out daily activities' worse quality of life and increased disability.

Cigarette smoking consider the most important risk factors air pollution, occupational chemicals and dusts, and frequent lower respiratory infections during childhood and not curable.

Symptom of COPD is the chronic and progressive shortness of breath which is most characteristic of the condition, wheezing, chest tightness and cough.

Thoracic hyperinﬂation caused by air trapping changes diaphragm muscle ﬁbers orientation in a zone of apposition (ZOA), which makes the contraction less eﬀective at lower rib cage expansion, The remodeling results in ﬂattening of the muscle and subsequent decreased diaphragmatic excursion

Osteopathic manipulative treatments (OMT) are hands-on manipulations of different body structures to increase systemic homeostasis and patient well-being include manipulation of the lymphatics, rib raising, diaphragmatic manipulations This treatment is used to stretch tight muscles, reduce pain, and improve circulation and lymphatic flow throughout the body

The diaphragmatic release technique is a manual technique that has beneficial effect on elongating tight diaphragmatic muscle fiber, improve perception of breathing assist in return doming shape to diaphragm, this lead to enhance pulmonary function, and to improve diaphragmatic mobility in both healthy individuals and patients with COPD

Rib raising is a manual technique increases thoracic mobility and lessens somatic dysfunctions of the area treated through normalized Parathoracic sympathetic ganglia.

The Thoracic Lymphatic Pumping Technique promote relaxation, facilitate blood flow and lymphatic drainage, reduce pain, normalize muscular tone and increase rib cage mobility .

this study aim to find out the effect of adding thoracic lymphatic pumping or rib raising manual techniques to diaphragmatic release in patients with COPD

This study will be conducted on 66 males of moderate to severe COPD patients. F tests - ANOVA: Fixed effects, omnibus, one-way F tests - ANOVA: Fixed effects, omnibus, one-way Analysis: A priori: Compute required sample size

Input:

Effect size f = 0.5 α err prob = 0.05 Power (1-β err prob) = 0.95 Number of groups = 3

Output:

Noncentrality parameter λ = 16,5000000 Critical F = 3,1428085 Numerator df = 2 Denominator df = 63 Total sample size = 66 Actual power = 0.9534748

ELIGIBILITY:
* include Stable COPD patients
* include Constant medication between the treatments.
* include Aged from 55TO 75 YEARS OLD
* include moderate to severe COPD
* include Smoker index <400
* exclude Rib or vertebral fracture
* exclude Skin disorder or scar in chest region or recent abdominal surgery.
* exclude Unwilling to complete in study
* exclude Cancer
* exclude Cognitive impairment to understand orders
* exclude severe osteoporosis
* exclude Smoker index >400

Ages: 55 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male gender with age 55 to70 years old stable copd
Enrollment: 66 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic Excursion | all assessment will be performed two times one pretreatment and will be repeated post treatment almost 2 months
  ultrasonography device applied on chest and used to measure the vertical movement of diaphragm
  unite of measure is centimeter (cm)
Level of Dyspnea | all assessment will be performed two times one pretreatment and then will be repeated post treatment almost 2 months
  Modified BORG Dyspnea Scale which measures level of dyspnea - Patients are asked "How much difficulty is your breathing?" and got a score 0 Nothing at all, 0.5 very very slight (just noticeable), 1 Very slight, 2 Slight, 3 Moderate, 4 Somewhat severe, 5 Severe, 7 Very severe, 9 Very, very severe (almost maximal), 10 Maximal.
Diaphragmatic thickness | all assessment will be performed two times one pretreatment and will be repeated post treatment almost 2 months
  ultrasonography device applied on chest and used to measure diaphragmatic thickness and change of flexibility of the diaphragm
  unite of measure is millimeter (mm)
Pulmonary function test (spirometry) | all assessment will be performed two times one pretreatment and will be repeated post treatment almost 2 months
  * patients will be asked to breathe in slowly and as deeply as possible, a breath out forcefully, then repeat 3 trials and will take the highest score during this will measure the following: Forced vital capacity (FVC) ,Forced expiratory volume first second (FEV1) as a percentage from predicted ,(FEV1/FVC) ratio ,Vital capacity (VC) ,Peak expiratory flow ,Forced expiratory flow 25%to75%
  * And ask patient to breath in and out as deep and fast as possible for 12 to 15 seconds to measure maximum voluntary ventilation
  unite of measurements: all measurements are taken as a percentage from predicted

CONTACTS AND LOCATIONS:
Overall Officials: SHERIN Hassan, PROF.DR., Principal Investigator — FACULTY OF PHYSICAL THERAPY Beni suef university
Locations (1):
- Faculty of Physical Therapy Beni Suef University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Spencer LM, Alison JA, McKeough ZJ. Do supervised weekly exercise programs maintain functional exercise capacity and quality of life, twelve months after pulmonary rehabilitation in COPD? BMC Pulm Med. 2007 May 16;7:7. doi: 10.1186/1471-2466-7-7. PMID 17506903
- [Result] Sleszynski SL, Kelso AF. Comparison of thoracic manipulation with incentive spirometry in preventing postoperative atelectasis. J Am Osteopath Assoc. 1993 Aug;93(8):834-8, 843-5. PMID 8407387
- [Result] Fei F, J Siegert R, Zhang X, Gao W, Koffman J. Symptom clusters, associated factors and health-related quality of life in patients with chronic obstructive pulmonary disease: A structural equation modelling analysis. J Clin Nurs. 2023 Jan;32(1-2):298-310. doi: 10.1111/jocn.16234. Epub 2022 Jan 30. PMID 35098602
- [Result] O'Donnell DE, Milne KM, James MD, de Torres JP, Neder JA. Dyspnea in COPD: New Mechanistic Insights and Management Implications. Adv Ther. 2020 Jan;37(1):41-60. doi: 10.1007/s12325-019-01128-9. Epub 2019 Oct 30. PMID 31673990
- [Result] Koch J, Tsui C, Talsma J, Pierce-Talsma S. Osteopathic Manipulative Treatment for Inhaled Rib Somatic Dysfunction. J Am Osteopath Assoc. 2020 Jul 28. doi: 10.7556/jaoa.2020.109. Online ahead of print. No abstract available. PMID 32722750
- [Result] Kaneko H, Shiranita S, Horie J, Hayashi S. Reduced Chest and Abdominal Wall Mobility and Their Relationship to Lung Function, Respiratory Muscle Strength, and Exercise Tolerance in Subjects With COPD. Respir Care. 2016 Nov;61(11):1472-1480. doi: 10.4187/respcare.04742. Epub 2016 Oct 18. PMID 27794081
- [Result] Marizeiro DF, Florencio ACL, Nunes ACL, Campos NG, Lima POP. Immediate effects of diaphragmatic myofascial release on the physical and functional outcomes in sedentary women: A randomized placebo-controlled trial. J Bodyw Mov Ther. 2018 Oct;22(4):924-929. doi: 10.1016/j.jbmt.2017.10.008. Epub 2017 Oct 25. PMID 30368336
- [Result] Halpin DM, Miravitlles M, Metzdorf N, Celli B. Impact and prevention of severe exacerbations of COPD: a review of the evidence. Int J Chron Obstruct Pulmon Dis. 2017 Oct 5;12:2891-2908. doi: 10.2147/COPD.S139470. eCollection 2017. PMID 29062228
- [Result] Global Initiative for chronic obstructive lung disease (GOLD).
- [Result] Ragab K. Elnaggar PhD & Mohammed A. Shendy Bulletin of Faculty of Physical Therapy
- [Result] Feizi H, Alizadeh M, Nejadghaderi SA, Noori M, Sullman MJM, Ahmadian Heris J, Kolahi AA, Collins GS, Safiri S. The burden of chronic obstructive pulmonary disease and its attributable risk factors in the Middle East and North Africa region, 1990-2019. Respir Res. 2022 Nov 19;23(1):319. doi: 10.1186/s12931-022-02242-z. PMID 36403049
- [Result] Bordoni B. Lymphatic Pump Manipulation in Patients with Chronic Obstructive Pulmonary Disease. Cureus. 2019 Mar 11;11(3):e4232. doi: 10.7759/cureus.4232. PMID 31123654